CLINICAL TRIAL: NCT06340399
Title: The Impact of Oral Branched-Chain Amino Acids Under Enhanced Recovery After Surgery on Reducing Postoperative Muscle Loss, Swallowing Difficulties, and Complications After Gastric Cancer Surgery: From Clinical to Precision Nutrition
Brief Title: BCAA in Patients Undergoing Gastric Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202312117RINE
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Perioeprative Muscle Loss

STUDY DESIGN:
Intervention Model Description: patients receiving BCAA
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: this is a open label use study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving BCAA (Experimental): patients undergoing BCAA before surgery to postoperative day 30
  Interventions: Dietary Supplement: BCAA
- patients not receiving BCAA (Placebo Comparator): patient not undergoing BCAA
  Interventions: Other: patient not administered BCAA

INTERVENTIONS:
Dietary Supplement: BCAA — patients administering BCAA
  Arms: patients receiving BCAA
Other: patient not administered BCAA — patients not administered BCAA
  Arms: patients not receiving BCAA

SUMMARY:
Older patients undergoing gastric cancer resection, at higher risk due to insufficient preoperative muscle mass, are more susceptible to SRML under surgical stress. This not only affects limb muscles but also impacts swallowing muscles, contributing to increased postoperative complications and mortality rates. Enhanced Recovery After Surgery (ERAS) has emerged as a multidisciplinary approach to facilitate postoperative recovery. This study aims to optimize oral nutrition under the ERAS model to observe its impact on SRML. BCAA is essential for skeletal muscles. However, there is limited research on the oral BCAA, whether before or after surgery, concerning SRML and its associated complications. The study entails an 18-month randomized controlled trial with 200 participants. One hundred individuals will take BCAA daily 5 to 14 days before surgery. After surgery, they can progress to a clear liquid diet around postoperative day five while continuing BCAA until 30 days postoperatively. The other one hundred participants will not receive BCAA. The study aims to investigate whether oral BCAA can reduce SRML, muscle loss, and decrease swallowing muscle strength, with observations on postoperative complications and outcomes within one year.

DETAILED DESCRIPTION:
Surgical Related Muscle Loss (SRML) is a prevalent complication following surgery, defined by a 10 percent or more reduction in muscle mass in at least one arm and one leg muscle by the seventh day postoperatively. Older patients undergoing gastric cancer resection, at higher risk due to insufficient preoperative muscle mass, are more susceptible to SRML under surgical stress. This not only affects limb muscles but also impacts swallowing muscles, contributing to increased postoperative complications and mortality rates. Enhanced Recovery After Surgery (ERAS) has emerged as a multidisciplinary approach to facilitate postoperative recovery. This study aims to optimize oral nutrition under the ERAS model to observe its impact on SRML. BCAA is essential for skeletal muscles. However, there is limited research on the oral BCAA, whether before or after surgery, concerning SRML and its associated complications.

The investigators entails an 18-month randomized controlled trial with 200 participants. One hundred individuals will take 3160 mg of BCAA daily 14 days before surgery. After surgery, they can progress to a clear liquid diet around postoperative day five while continuing BCAA until 30 days postoperatively. The other one hundred participants will not receive BCAA. The study aims to investigate whether oral BCAA can reduce SRML, muscle loss, and decrease swallowing muscle strength, with observations on postoperative complications and outcomes within one year.

Regarding the swallowing measurement, high-resolution impedance manometry, the most accurate tool for assessing swallowing muscle strength, will be used. The ultrasound will also be used to investiagte the muscle loss. We will also investigate the genome associated BCAA study.

ELIGIBILITY:
Inclusion Criteria:

* I) Patients confirmed to have gastric adenocarcinoma (one type of stomach cancer) through endoscopic biopsy prior to surgery, with the selection based on this type representing the majority of gastric cancer cases at National Taiwan University Hospital.

II) Patients aged between 20 and 90, irrespective of gender, are eligible for inclusion.

III) Severity of gastric cancer: Patients with clinical stages I to III and no distant metastasis, undergoing complete tumor resection, according to the 15th edition of the Japanese Gastric Cancer Classification.

IV) Postoperative status assessment of patients: Utilizing the Eastern Cooperative Oncology Group (ECOG) scoring system to assess the performance status of cancer patients. Scores of 0-2 indicate relatively good overall health, normal daily activities, and the ability to tolerate cancer-related treatments.

V) Patients with normal general blood biochemistry values, including Aspartate Aminotransferase (AST), Alanine aminotransferase (ALT), Total Bilirubin, and Creatinine.

VI) Patients provide written informed consent prior to participation.

Exclusion Criteria:

- I) Exclusion criteria include patients with other diseases and complications such as: concurrent cancers in the stomach, the need for additional surgeries due to postoperative complications or unstable conditions, heart diseases categorized as New York Heart Association functional class ≥2 with thrombotic conditions, lung diseases categorized as Hugh-Jones grade ≥4, and patients currently undergoing insulin therapy.

II) Patients taking preventive medication for gastric cancer, such as those undergoing treatment for Helicobacter pylori infection.

III) As this study involves preoperative and postoperative rehabilitation exercises, patients with impaired physical function are not suitable.

IV) Individuals allergic to eggs, soybeans, or thiamine.

V) Patients already supplementing with BCAA (branched-chain amino acids).

VI) Individuals with psychological disorders that may affect their ability to provide informed consent or adhere to the study protocol.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the occurrence of surgical related muscle loss | before surgery to postoperative day 7
  examined the surgical related muscle loss occurence

IPD SHARING:
Plan to Share IPD: No
due to ethical issue